CLINICAL TRIAL: NCT04643054
Title: Efficacy and Safety of Ovotransferrin in COVID-19 Patients With Mild-to-Moderate Disease
Brief Title: Efficacy and Safety of Ovotransferrin in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Antonio Cascio, Chief Infectious and Tropical Diseases Departmemt, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201116
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: Ovotransferrin
MeSH Terms: conditions — COVID-19 | interventions — Conalbumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ovotransferrin (Experimental): Dietary Supplement: Ovotransferrin
  Interventions: Dietary Supplement: Ovotransferrin
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Ovotransferrin — Administering 200 mg of ovotransferrin orally in addition to the standard of care therapy for 10 days
  Arms: Ovotransferrin

SUMMARY:
Chicken egg consists of three main components, egg white (56%), yolk (33%) and shell (11%). The key component of egg white is 88 percent water and 12 percent solids, of which over 90 percent are protein. Ovalbumin, ovotransferrin, and ovomucoid are considered the main proteins, while ovomucin, lysozyme, ovoglobulin, ovomacroglobulin, ovoglycoprotein, ovoflavoprotein, thiamin-binding proteins, ficin/papain inhibitors, avidin, and cystatin are the minor white proteins of the embryo. These proteins and their peptides have been recognized as antioxidants, antimicrobials, metal-chelators, anti-viral, anti-tumor, and angiotensin-converting enzyme (ACE)-inhibitors for their functional significance SARS-CoV-2 virus activates the human cell ACE2 receptor, triggering a series of deleterious events. In COVID19, renin-angiotensin is upregulated and the pathway is overexpressed and a progressive cytokine storm is always observed. In all these pathogenic processes, ovotransferrin could play a modifier function to enhance the condition. Ovotransferrin can be beneficial to the antioxidant effects of Angiotensin II by inhibiting NF-kB. Ovotransferrin is an immunomodulator that downregulates pro-inflammatory cytokines including TNF-α, IL-6, and IL-1 that could extinguish the cytokine storm. Ovotransferrin can also serve as a protective agent against COVID19 cardiotoxicity due to disruption in the ACE2-mediated signaling pathway, cytokine storm, pulmonary dysfunction, and side effects of medications.

In patients with coronavirus infection, provided ovotransferrin's possible protective effects, it is suggested as a supportive and therapeutic alternative.

Given this background, in the light of the current COVID-19 emergency, it is the intention of the investigators to conduct a prospective, randomized, open-label, controlled study in the cohort of hospitalized patients with covid-19 pneumonia, administering 200 mg of ovotransferrin orally in addition to the standard of care therapy (SOC).

The investigators hypothesize that the use of ovotransferrin will be associated with an earlier improvement of clinical and humoral parameters after 10 days of ovotransferrin treatment when compared to the group of patients provided with standard care.

DETAILED DESCRIPTION:
Chicken egg consists of three main components, egg white (56%), yolk (33%), and shell (11%). The key component of egg white is 88 percent water and 12 percent solids, of which over 90 percent are protein. Ovalbumin, ovotransferrin, and ovomucoid are considered the main proteins, while ovomucin, lysozyme, ovoglobulin, ovomacroglobulin, ovoglycoprotein, ovoflavoprotein, thiamin-binding proteins, ficin/papain inhibitors, avidin, and cystatin are the minor white proteins of the embryo. These proteins and their peptides have been recognized as antioxidants, antimicrobials, metal-chelators, anti-viral, anti-tumor, and angiotensin-converting enzyme (ACE)-inhibitors for their functional significance. Among these functional properties, the antioxidant ability is essential to food processing. Generation of reactive oxygen species (ROS) and free radicals is an integral part of biological processes affecting all living organisms in energy production. Ovotransferrin (OTf), which constitutes 12% of the total white egg protein, is known as an iron binder and transporter in animals and can thus be used as an iron replacement, antimicrobial or antioxidant. Japanese researchers find ovotransferrin in a redox-dependent method generates observable self-cleaning.

OTf is composed of 686 amino acids and has a molecular mass of 77.90 kDa. It is a superoxide dismutase (SOD)-mimicking protein with a potent superoxide anion (O2 _-)-scavenging activity and showed dramatically higher scavenging activity than some known antioxidants, such as serum albumin or ascorbate. Interestingly, metal-bound OTfs such as Fe2+-OTf, Mn2+-OTf, Cu2+-OTf exhibited greater O2 _- dismutation capacity than the apoprotein. Conjugation of OTf with small molecules such as catechin shows improved antioxidant activity. During in vitro experiments, OTf displayed some antioxidant effects and its hydrolysates showed approximately 3,2 to 13,5 times higher superoxide anion scavenging activity and better copper/calcium scavenging activity than OTf. Furthermore, autocleaved OTf showed higher antioxidant activity than the natural OTf, and the hydrolysates of autocleaved OTf showed stronger antioxidant activity than those of the autocleaved one.

The peptide IRW, resulting from hydrolysis, exhibited a high-oxygen radical-scavenging that could be related to tryptophan. In addition, two high antioxidant activity tetrapeptides (WNIP and GWNI) were found in OTf thermolysin digests. WNI's motif seemed to be responsible for the high antioxidant potential as amino acid residues coupled with both peptides' N or C terminus decreased their antioxidant capacity. Moreover, when tested in endothelial cells, the peptide GWNI showed the ability to reduce reactive oxygen species generation. Other antioxidant peptides previously reported from OTf using the oxygen radical absorbance ability, on the other hand showed no antioxidant activity in cells, showed deficiencies in cell-free in vitro methods for antioxidant studies, and highlighted the need to use more biological systems such as culture cells to test antioxidant peptides. OTf-derived hydrolyzates obtained with HCl at pH 2.5 or other enzymes such as protamex, alkalase, trypsin, neutrase, flavorzyme, maxazyme, collupulin, protex, promod 278 and alpha-chymotrypsin showing higher superoxide anion scavenging activity and radical oxygen absorption ability than intact protein and showing protective effects against oxidative stress-induced DNA.

Due to their anti-inflammatory and antioxidant properties, otrf-derived peptides, including IRW, IQW, and KVREGT, are viable treatment agents for endothelial dysfunction and CVD prevention. They de-regulate the expression of the cytokine-induced inflammatory protein in the vascular endothelium by modulating the pathway NF-μB. Recent research also revealed that KVREGT has a significant role to inhibit ACE and promote vasodilation. IQW impedes ACE, promoting antioxidation.

Ovotransferrin and lactoferrin are iron-binding proteins with natural immunity-related antiviral and antibacterial activities, displaying marked sequence and structural homologies. Two hen ovotransferrin fragments DQKDEYELL (hOtrf219-227) and KDLLFK (hOtrf269-301 and hOtrf633-638) have registered antiviral activity against Marek virus infection of chicken embryo fibroblasts. These fragments have sequence homology with two bovine lactoferrin fragments with antiviral activity towards herpes simplex virus, indicating that these fragments may play a role in exploiting intact protein antiviral activity towards herpes viruses. NMR analysis showed that these chemically synthesized peptides had no favorite solution conformation, suggesting that both the amino acid sequence and the conformation in the intact protein are necessary for antiviral action.

SARS-CoV-2 virus activates the human cell ACE2 receptor, triggering a series of deleterious events. In COVID19, renin-angiotensin is upregulated and the pathway is overexpressed and a progressive cytokine storm is always observed. In all these pathogenic processes, ovotransferrin could play a modifier function to enhance the condition. Ovotransferrin can be beneficial to the antioxidant effects of Angiotensin II by inhibiting NF-kB. Ovotransferrin is an immunomodulator that downregulates pro-inflammatory cytokines including TNF-α, IL-6, and IL-1 that could extinguish the cytokine storm. Ovotransferrin can also serve as a protective agent against COVID19 cardiotoxicity due to disruption in the ACE2-mediated signaling pathway, cytokine storm, pulmonary dysfunction, and side effects of medications.

In patients with coronavirus infection, provided ovotransferrin's possible protective effects, it is suggested as a supportive and therapeutic alternative.

Given this background, in the light of the current COVID-19 emergency, it is the intention of the investigators to conduct a prospective, randomized, open-label, controlled study in the cohort of hospitalized patients with covid-19 pneumonia, administering 200 mg of ovotransferrin orally in addition to the standard of care therapy (SOC).

The investigators hypothesize that the use of ovotransferrin will be associated with an earlier improvement of clinical and humoral parameters after 10 days of ovotransferrin treatment when compared to the group of patients provided with standard care.

ELIGIBILITY:
Inclusion Criteria:

* Positive swab test of SARS-CoV-2
* Pneumonia related to SARS-CoV-2
* Signature of informed consent
* Absence of allergies to egg proteins

Exclusion Criteria:

* Unsigned informed consent
* Negative swab test of SARS-CoV-2
* Allergy to egg proteins
* Pregnancy and breastfeeding
* Mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 48hours
  Change of hospital mortality

SECONDARY OUTCOMES:
C reactive protein (CRP) levels | 48 hours
  Reduction of CRP levels > 50% in comparison with CRP levels at the admission, within 48 hours after the administration
IL-6 levels | 48 hours
  Reduction of IL-6 levels > 50% in comparison with IL-6 at the admission, within 48 hours after the administration
D-dimer levels | 48 hours
  Reduction of D-dimer levels > 50% in comparison with D-dimer at the admission, within 48 hours after the administration
Hospital stay | up to 24 weeks
  Length of hospital stay
Duration of positive PCR swab | 5 days
  Time length of negativization of PCR molecular swab

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cascio, MD, PhD, Principal Investigator — AOU Policlinico "P. Giaccone" - University of Palermo, Italy
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abeyrathne EDNS, Huang X, Ahn DU. Antioxidant, angiotensin-converting enzyme inhibitory activity and other functional properties of egg white proteins and their derived peptides - A review. Poult Sci. 2018 Apr 1;97(4):1462-1468. doi: 10.3382/ps/pex399. PMID 29340654
- [Background] Benede S, Molina E. Chicken Egg Proteins and Derived Peptides with Antioxidant Properties. Foods. 2020 Jun 3;9(6):735. doi: 10.3390/foods9060735. PMID 32503187
- [Background] Chen S, Jiang H, Peng H, Wu X, Fang J. The Utility of Ovotransferrin and Ovotransferrin-Derived Peptides as Possible Candidates in the Clinical Treatment of Cardiovascular Diseases. Oxid Med Cell Longev. 2017;2017:6504518. doi: 10.1155/2017/6504518. Epub 2017 Mar 13. PMID 28386310
- [Background] Giansanti F, Massucci MT, Giardi MF, Nozza F, Pulsinelli E, Nicolini C, Botti D, Antonini G. Antiviral activity of ovotransferrin derived peptides. Biochem Biophys Res Commun. 2005 May 27;331(1):69-73. doi: 10.1016/j.bbrc.2005.03.125. PMID 15845359